CLINICAL TRIAL: NCT04172129
Title: Assessment of Implant Fixation and SF-36 for Short Hip-Stems - A Prospective Clinical Study
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: R11014-3-D
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Primary and Secondary Coxarthrosis; Dysplasia Coxarthrosis; Post-traumatic Necrosis of the Femoral Head
Keywords: Nanos; THA; MBRSA
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NANOS: NANOS™ Neck Preserving Hip Stem
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty

SUMMARY:
The primary purpose of this study was to evaluate the implant fixation of the NANOS™ Neck Preserving Hip Stem (OHST Medizintechnik AG, distributed by Smith & Nephew GmbH, Marl, Germany) by measuring the migration of the implant using the model-based roentgen stereophotogrammetric analysis (MBRSA).

ELIGIBILITY:
Inclusion Criteria:

* Subject required primary total hip arthroplasty unilateral or bilateral with a diagnosis of primary and secondary coxarthrosis, dysplasia coxarthrosis and post-traumatic necrosis of the femoral head confirmed by x-ray analysis. For bilateral subjects at least three months between surgical procedures were required.
* Subject was willing to consent to participate in the study and planned to be available for the follow-up examinations.
* Subject had normal motor function of the lower extremities, documented through clinical examinations and lack of signs of a neurological disease with changed motor function.
* Subject was 30 to 65 (inclusive) years of age at time of surgery.

Exclusion Criteria:

* Subject had previous bone or soft tissue surgery of the affected hip except for arthroscopic surgery.
* Subject had a local or systemic infection.
* Subject had previously diagnosed osteoporosis.
* Subject had a femoral neck angle of >145°.
* Subject had a femoral neck angle of <125°.
* Subject had a disease of the cardiovascular system involving particularly reduced load capacity in the everyday life, counting as contraindication of physical stress (American Society of Anaesthesiologists' (ASA) Score 3 or 4).
* Subject had a documented allergy against elements of the implanted device.
* Subject had a neurological disease with changed motor function.
* Subject was pregnant.
* Subject had a Body Mass Index (BMI) > 30.
* Subject suffered from alcoholism or addictive disorders.
* Subject needed a revision hip arthroplasty.
* Subject had an insufficient command of the language to understand patient information and consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified in the primary care clinic with need for total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-04-26 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of migration pattern of the Nanos stem | 2 years
  Measuring migration used the model-based RSA method
Change in quality of life | 2 years
  Measuring change in quality of life using the Short Form (SF) 36 Mental Component Score
  * Minimum Value: 0 (worst outcome)
  * Maximum Value: 100 (best outcome)

SECONDARY OUTCOMES:
Harris Hip Score | 2 years
  Investigator assessed outcome score Minimum: 0 (worst outcome) Maximum: 100 (best outcome)
University of California, Los Angeles (UCLA) scale | 2 years
  Score rating the patient's current activity level
  * Minimum: 1 (wholly inactive subject)
  * Maximum: 10 (totally active subject)
Pain Visual Analogue Scale | 2 years
  Score representing patient's current pain intensity
  * Minimum: 0 (no pain)
  * Maximum: 100 (very severe pain)
Postel Merle d'Aubigné-Score | 2 years
  Score grading the functional value of the hip
  * Minimum: 0 (worst outcome)
  * Maximum: 6 ( best outcome)
  Grading is done in each of the three dimensions: pain, mobility and ability to walk.
Hip Disability and Ostheoarthritis Outcome Score | 2 years
  Patient reported outcome
  * Minimum: 0 (best outcome)
  * Maximum: 96 (worst outcome)
Radiographic Evaluation | 2 years
  Evaluation of radiographic images regarding implant position, implant fixation, heterotopic ossifications (HO), radiolucencies, osteolysis, atrophy and hypertrophy
Number of adverse events | 2 years
  Collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Henning Windhagen, Prof. Dr. med., Principal Investigator — Orthopädische Klinik der Medizinischen Hochschule Hannover
Locations (1):
- Orthopädische Klinik der Medizinischen Hochschule Hannover, Hanover, Germany